CLINICAL TRIAL: NCT01493752
Title: Investigation of the Effect of Dietary Nitrate Treatment on Endothelial Function, Platelet Reactivity in Hypercholesterolemics Without Known Cardiovascular Disease or Atherosclerosis.
Brief Title: Investigation of the Effect of Dietary Nitrate Treatment on Endothelial Function and Platelet Reactivity in Hypercholesterolemics.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Principal Investigator, Amrita Ahluwalia, Professor of Vascular Pharmacology, Queen Mary University of London
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: 11/LO/0715
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate-rich beetroot juice (Active Comparator): Six weeks once daily dose of nitrate rich beetroot juice
  Interventions: Dietary Supplement: beetroot juice
- Nitrate deplete beetroot juice (Placebo Comparator): six weeks daily dose beetroot juice (nitrate deplete)
  Interventions: Dietary Supplement: beetroot juice

INTERVENTIONS:
Dietary Supplement: beetroot juice — 250mls daily beetroot juice

SUMMARY:
Diets rich in fruit and vegetables reduce the risk of strokes and heart attacks, however the exact cause of this beneficial effect is uncertain. Evidence suggests that certain vegetables, including beetroot and the green leafy vegetables, possess high inorganic nitrate concentrations. The investigators recent evidence suggests that inorganic nitrate provides a source of gas called nitric oxide in the body that exerts a number of beneficial effects upon the heart and blood vessels . The investigators have previously shown that beetroot juice ingestion improves blood vessel (vascular endothelial) and platelet function in healthy volunteers. Studies by the investigators show that these effects are due to conversion of nitrate to nitrite by symbiotic (helpful) bacteria (located on the tongue) and subsequent conversion of nitrite to nitric oxide in blood vessels. The investigators now wish to explore whether dietary nitrate, via its beneficial effects on platelets and blood vessels, might improve indices of atherosclerotic disease progression in high risk individuals (hypercholesterolemics). Recruits will have high cholesterol and no known atherosclerosis and will not yet be on any anti-cholesterol medications. Volunteers will consume a daily dose of beetroot juice or placebo nitrate-free juice for six weeks. Vascular function will be assessed using non-invasive techniques at the beginning and at the end of the study using ultrasound measurement of flow mediated dilatation (FMD) of the brachial artery in the arm and pulse wave analysis (PWA) and pulse wave velocity (PWV) to measure arterial compliance. To assess impact on platelet function, blood samples will also be taken at the start and at the end of the study.

DETAILED DESCRIPTION:
Please refer to brief summary.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be between 18-80 years of age.
2. They will be largely newly diagnosed patients with hypercholesterolemia (total serum cholesterol>6.0mmol/L or any elevation of total cholesterol, LDL cholesterol or triglycerides with a QRISK 2 score >15%).
3. We will include patients with familial hypercholesterolemia. These patients in general will either be managed in primary care alone or will attend the clinic following referral from general practitioners for further investigation following routine health tests.
4. In addition, patients who have been referred due to inability to tolerate statin treatment will be included.
5. They will be recruited into the study if they are interested in taking part in research, do not have any exclusion criteria on screening and give their written informed consent.

Hypercholesterolemics will be screened by taking a medical history and physical examination, blood pressure measurement and urine sample taken to check for diabetes. The subject will continue his/her usual diet and exercise regime prior to diagnosis of hypercholesterolemia for purposes of this study. They will not be taking any additional vitamin or food supplements for the duration of the study.

Exclusion criteria

1. A history of symptomatic ischemic heart disease (angina, previous myocardial infarction, acute coronary syndrome) or other known atherosclerosis.
2. A history of heart failure NYHA class 2-4 or severe LV dysfunction LVEF<30% regardless of symptom status.
3. Use of statins within 2 months of screening visit.
4. A history of diabetes.
5. Systemic autoimmune disease such as rheumatoid arthritis, connective tissue disease, or other conditions known to be associated with chronic inflammation such as inflammatory bowel disease.
6. Any use of non steroidal anti-Inflammatory drugs, antiplatelet agents or steroids within two months of commencing study or likely future use required during the study.
7. Subjects with any acute infection, or significant trauma (burns, fractures).
8. Subjects who have donated > 500mls blood within 56 days prior to study medication administration.
9. Anaemia with Hb <10g/dl, or any other known blood disorder or significant illness that may affect platelet function, and coagulation. Known essential hypertension on antihypertensive medication is not a contraindication.
10. History of malignancy within the past 5 years other than non-melanoma skin cancer.
11. Any current life threatening condition including severe chronic obstructive airways disease, HIV infection, life threatening arrhythmia that may prevent subject completing the study.
12. Alcohol/drug abuse within the past 6 months of screening visit.
13. Excess alcohol consumption as defined as regular weekly consumption of >28 units male and >21 units female. (Department of Health Guidelines)
14. Use of an investigational device or investigational drug within 30 days or 5 half lives (whichever is longer) preceding the first dose of study medication.
15. Any non stable dosing of ongoing medication regimens throughout the study trial.
16. A history of chronic viral hepatitis (including presence of hepatitis B surface antigen or hepatitis C antibody or other chronic hepatic disorder.)
17. Abnormal liver function due to acute or chronic liver conditions 3 x upper limit of normal at screening.
18. Renal impairment with creatinine clearance (eGFR) of <50ml/min at screening.
19. Pregnancy at time of screening or intention of getting pregnant during course of study.
20. Current smokers or ex smokers who stopped smoking <3 months prior to administration of study medication.
21. BMI <18.5 or > or = 40kg/m2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Flow Mediated Dilatation (FMD) | 6 weeks
  Brachial artery ultrasound FMD as a measure of endothelial function before and after beetroot juice

SECONDARY OUTCOMES:
Platelet aggregation studies, pulse wave analysis, pulse wave velocity, plasma nitrate and nitrate concentration. | after 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Barts & The London Medical School, William Harvey Research Institute, London, United Kingdom

REFERENCES:
- [Derived] Velmurugan S, Gan JM, Rathod KS, Khambata RS, Ghosh SM, Hartley A, Van Eijl S, Sagi-Kiss V, Chowdhury TA, Curtis M, Kuhnle GG, Wade WG, Ahluwalia A. Dietary nitrate improves vascular function in patients with hypercholesterolemia: a randomized, double-blind, placebo-controlled study. Am J Clin Nutr. 2016 Jan;103(1):25-38. doi: 10.3945/ajcn.115.116244. Epub 2015 Nov 25. PMID 26607938